CLINICAL TRIAL: NCT07262970
Title: Intermediate-Size Cohort EAP for Ersodetug in Patients With Refractory Hypoglycemia Due to Tumor-Associated Hyperinsulinism (Tumor HI) Who Are Unable to Participate in a Clinical Trial
Brief Title: Intermediate-Size Cohort EAP for Ersodetug in Patients With Inadequately Controlled Hypoglycemia Related to a Tumor
Status: Available | Type: Expanded Access
Sponsor: Rezolute (Other)
Responsible Party: Sponsor
Other Study IDs: RZ358-303
Record Dates: First submitted 2025-11-21; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Tumor-associated Hyperinsulinism (Tumor HI)
Keywords: Insulinoma; Islet cell tumor (ICT); Ectopic insulinoma; Extra-pancreatic insulinoma; Pro-insulinoma; Non-islet cell tumor hypoglycemia (NICTH); Non Islet Cell Tumor; IGF 2 mediated non islet cell tumor hypoglycemia; IGF-oma, IGF-2-oma, Big IGF-2-oma; IGF-2, Big IGF-2; Neuroendocrine tumor (NET); PNET; Hypoglycemia; Paraneoplastic; Tumor/cancer associated hypoglycemia; Tumor/cancer induced hypoglycemia; Tumor/cancer mediated hypoglycemia; Hypoglycemia due to tumor/cancer; Doege-Potter Syndrome; Paraneoplastic hypoglycemia; Hyperinsulinemia; IGF-2 mediated hypoglycemia; HCC; Liposarcoma; Fibrosarcoma; Hypoglycemia due to HCC; Hypoglycemia due to liposarcoma; Hypoglycemia due to fibrosarcoma; Clinical Trials for: -Insulinoma -proinsulinoma -extrapancreatic insulinoma -non-islet cell tumor -IGF-oma -HCC -Liposarcoma -Fibrosarcoma; Expanded Access; Cohort Expanded Access; EAP; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Insulinoma; Adenoma, Islet Cell; Neuroendocrine Tumors; Neuroectodermal Tumors, Primitive; Hypoglycemia; Neoplasms; Hyperinsulinism; Liposarcoma; Fibrosarcoma

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Ersodetug (9 mg/kg) + SOC — Open-Label Participants with a diagnosis of Tumor HI (insulin- or IGF-producing tumors)

SUMMARY:
This expanded access program is intended to provide ersodetug, an investigational drug, to eligible participants who suffer from inadequately controlled hypoglycemia due to tumor-associated hyperinsulinism and are unable to participate in ersodetug clinical trial. Participation is open to participants who meet the eligibility criteria and for whom access to the investigational drug is deemed appropriate by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled hypoglycemia due to documented tumor HI (including but not limited to: insulin/pro-insulin producing pancreatic/non-pancreatic neuroendocrine tumors, insulin-like growth factor-producing NICTH) that is not adequately managed with available SoC anti-hypoglycemic therapies (per Treating Physician's judgement).
* Inability to participate in any ersodetug clinical trial.
* Women of childbearing potential (WOCBP) must not be pregnant or breast feeding, and must be willing to use effective contraceptive measures or practice complete sexual abstinence to prevent pregnancy for the duration of the Cohort EAP AND for at least 5 months after receiving the last dose of ersodetug.
* Male participants with female partner of childbearing potential must be willing to use effective contraceptive measures or practice complete sexual abstinence to prevent pregnancy for the duration of the Cohort EAP AND for at least 5 months after receiving the last dose of ersodetug.

Exclusion Criteria:

* Any unexplained out-of-range laboratory value (other than glucose) that is assessed as clinically significant impacting patient safety if enrolled by the Treating Physician. Laboratory or other abnormalities that are considered related to the underlying disease or associated therapies that do not pose additional safety risk for participation per Treating Physician may be allowed upon Medical Monitor approval.
* Evidence of active infection including (but not limited to) human immunodeficiency virus, hepatitis B, or hepatitis C.
* Known allergy or sensitivity to ersodetug or any component of the drug.
* Treatment with an investigational drug or device within 30 days or 5 t½ of the investigational drug before the planned 1st dose of ersodetug, whichever is longer. However, if the Treating Physician and Medical Monitor consider no significant risk of drug-drug interaction and potential benefit to outweigh the risk, then the participant may be allowed to participate. Participation in registries and/or purely diagnostic studies are allowed.
* Any organ condition, concomitant disease (including but not limited to any psychiatric illness, severe alcoholism, or drug abuse, cardiac, hepatic, or kidney disease), or other abnormality that itself, or the treatment of which, could interfere with the conduct of the program (e.g., may affect absorption, distribution, metabolism, or elimination of the program drug) or that, in the opinion of the Treating Physician and/or Medical Monitor would pose an unacceptable risk to the participant in the program.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult